CLINICAL TRIAL: NCT05724589
Title: The Effectiveness of Epidermal Growth Factor Serum for the Improvement of Facial Skin Hydration, Elasticity, Pigmentation, and Wrinkles at the Institute of Dermatology: a Single-centered Pilot Study With a One-group Before-and-after Design
Brief Title: The Effectiveness of Epidermal Growth Factor Serum in Improve Facial Skin Hydration, Elasticity, Pigmentation, and Wrinkles.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Dermatology, Thailand (Other Government)
Responsible Party: Principal Investigator, Supawee Phanmamuang, MD, Resident of Dermatology, Institute of Dermatology, Thailand
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 008/2565
Record Dates: First submitted 2023-01-30; First posted 2023-02-13 (Actual); Results first posted 2025-07-31 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Aging
MeSH Terms: interventions — Epidermal Growth Factor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Epidermal Growth Factor Serum Application (Experimental): Participants received Epidermal growth factor serum application on the face daily for two months compared to pre and post-results of skin quality.
  Interventions: Drug: Epidermal Growth Factor

INTERVENTIONS:
Drug: Epidermal Growth Factor — Apply facial twice daily.
  Other Names: Epidermal Growth Factor Serum

SUMMARY:
EGF is a polypeptide that promotes cell differentiation and collagen production while decreasing melanin production. This study is designed to study its effectiveness in improving the texture and appearance of facial skin after daily topical application. We hypothesized that EGF would improve facial skin hydration, elasticity, pigmentation, and wrinkles.

DETAILED DESCRIPTION:
All patients gave written informed consent for epidermal growth factor serum application on the face. The pilot study enrolls thirty patients compared to pre and post-serum used to evaluate facial skin hydration, transepidermal water loss, elasticity, pigmentation, and wrinkles measured by corneometer, tewameter, cutometer, visioscan, and mexameter respectively on day 0, then 8, 12, and 16 weeks. The study evaluates subject satisfaction and side effects after serum application as secondary outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Thai
* Mild to moderate facial skin condition, as measured by 1-2 points on the hyperpigmentation status scale or 2-3 points on the wrinkle severity grading scale.

Exclusion Criteria:

* Use of lotions or skin care products containing ingredients such as vitamin A/C, hydroquinone, or anti-aging agents.
* Sunbathing
* Hypersensitivity to serum components
* Pregnancy and breast-feeding
* Active skin diseases such as eczema or atopic dermatitis at the application site

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2023-01-30 (Actual); Primary Completion 2024-06-05 (Actual); Study Completion 2024-12-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chumsaeng Chumsaengsri, Principal Investigator — Institute of Dermatology
Locations (1):
- Institute of Dermatology, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Pre-assignment Details of 28 enrolled participants, all met inclusion criteria.
Units Other Than Participants: face
Period: Overall Study
Arm/Group | Epidermal Growth Factor Serum Application
Started | 28; 28 face
Completed | 27; 27 face
Not Completed | 1; 1 face
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Population: Twenty-eight patients participated in a pilot study. The study involved pre- and post-serum assessments at four different time points (0, 8, 12, and 16 weeks). Various instruments, including tewameter, corneometer, cutometer, mexameter, and visioscan, were used for measurements.
Units Other Than Participants: face
Arm/Group | Epidermal Growth Factor Serum Application
Number analyzed (Participants) | 28
Number analyzed (face) | 28
Age, Continuous [Mean (Standard Deviation); unit: ัyears] | 52 (8.41)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 28
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 28
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Thailand | 28
Underlying disease [Count of Participants; unit: Participants]
  Hypertension | 4
  Diabetes | 2
  Other | 3
  No | 18
  No identify. | 1
Occupation [Count of Participants; unit: Participants]
  Government employee | 1
  Permanent employee | 3
  Temporary employee | 14
  Security guard | 4
  Government officer | 1
  Office worker | 4
  No identify. | 1
Fitzpatrick skin type [Count of Participants; unit: Participants] — Participants were classified using the Fitzpatrick Skin Type Scale, which ranges from Type I (very fair skin, always burns, never tans) to Type VI (deeply pigmented skin, never burns). Classification was based on self-reported skin response to sun exposure and visual assessment. In this study, Types I-II were considered more sensitive to treatment-related skin reactions (worse outcomes), while Types V-VI, with higher melanin levels, were considered less prone to visible reactions (better outcomes).
  Participants
    III | 5
    IV | 23
Hormone use [Count of Participants; unit: Participants]
  No | 27
  Yes | 1
Pregnancy [Count of Participants; unit: Participants]
  No | 28
  Yes | 0
Menopause [Count of Participants; unit: Participants]
  No | 18
  Yes | 10
Smoking [Count of Participants; unit: Participants]
  No | 28
  Yes | 0
Alcohol drinking [Count of Participants; unit: Participants]
  No | 27
  Yes | 1
Regular sun expose [Count of Participants; unit: Participants]
  No | 28
  Yes | 0

OUTCOME MEASURES:

1. Primary Outcome: Facial Skin Hydration
Description: Facial skin hydration was measured using a Corneometer, which provides readings in arbitrary units (a.u.). Measurements were taken at baseline (Day 0), Week 8, Week 12, and Week 16 under standardized environmental and procedural conditions to ensure reliability and accuracy. Higher values indicate better skin hydration, while lower values indicate increased dryness.
Time Frame: 4 months (Baseline, Week 8, Week 12, Week 16)
Population: The analysis population included 28 subjects initially recruited for this study. Participants were assessed at four time points: baseline (Day 0), Week 8, Week 12, and Week 16. One participant was lost to follow-up after Week 12 and Week 16.
Measure: Mean (Standard Deviation); unit: arbitrary units
Units Other Than Participants: face
Arm/Group | Epidermal Growth Factor Serum Application
Number analyzed (Participants) | 28
Number analyzed (face) | 28
arbitrary units
  Baseline | 56.043 (1.900)
  8 weeks | 58.300 (1.567)
  12 weeks: number analyzed (Participants) | 27
  12 weeks: number analyzed (face) | 27
  12 weeks | 55.852 (1.583)
  16 weeks: number analyzed (Participants) | 27
  16 weeks: number analyzed (face) | 27
  16 weeks | 58.714 (1.568)
Statistical Analysis 1: Comparison: Epidermal Growth Factor Serum Application; Skin hydration was evaluated longitudinally using repeated measures ANOVA at Baseline, Week 8, Week 12, and Week 16. This pre-specified statistical test assessed within-subject changes over time to determine the efficacy of the serum; Test type: Superiority — A repeated measures ANOVA was selected to analyze changes in skin hydration across four time points within the same participants; p = 1.000, ANOVA — The p-value reflects the overall test for difference in hydration over time and is not adjusted for multiple comparisons. The pre-defined threshold for statistical significance was p < 0.05; No additional adjustments were applied. Degrees of freedom and sphericity assumptions were checked; Mean Difference (Final Values) = 2.671 — The mean difference was calculated based on changes in skin hydration from baseline to Week 16 using repeated measures ANOVA, in accordance with the pre-specified statistical analysis plan; The overall p-value corresponds to the repeated measures ANOVA evaluating changes over four time points. No multiplicity adjustments were applied

2. Primary Outcome: Transepidermal Water Loss
Description: measured by tewameter on day 0, then at 8, 12, and 16 weeks.
Time Frame: 4 months
Population: The analysis population for this study on Transepidermal Water Loss (TEWL) utilizing Tewameter measurements comprised a total of 28 initially recruited subjects. These participants were assessed at four distinct time points: day 0 (baseline), 8 weeks, 12 weeks, and 16 weeks. One subject loss follow-up at week 12 and week 16.
Measure: Mean (Standard Deviation); unit: g/m²·h
Units Other Than Participants: face
Arm/Group | Epidermal Growth Factor Serum Application
Number analyzed (Participants) | 28
Number analyzed (face) | 28
g/m²·h
  Baseline | 11.815 (1.221)
  8 weeks | 8.761 (0.623)
  12 weeks: number analyzed (Participants) | 27
  12 weeks: number analyzed (face) | 27
  12 weeks | 8.400 (0.516)
  16 weeks: number analyzed (Participants) | 27
  16 weeks: number analyzed (face) | 27
  16 weeks | 8.160 (0.559)
Statistical Analysis 1: Comparison: Epidermal Growth Factor Serum Application; Test type: Superiority — The statistical analysis in this study to assess changes in Transepidermal Water Loss (TEWL) after serum application involved a repeated measures analysis of variance (ANOVA). This approach allows for the examination of differences in TEWL across multiple time points (baseline, 8 weeks, 12 weeks, and 16 weeks) within the same individuals. The use of repeated measures ANOVA accounts for the correlated nature of the data, as multiple measurements are obtained from each participant over time; p = 0.096, ANOVA — A repeated measures ANOVA was used to assess changes in hydration over time. The mean difference between baseline and 16 weeks was -3.656 (arbitrary units). Results are presented in the corresponding outcome measure table; Mean Difference (Final Values) = -3.656

3. Primary Outcome: Facial Skin Elasticity (R2 Parameter Via Cutometer)
Description: Skin elasticity was assessed using a Cutometer with the R2 parameter (Ua/Uf), which measures gross elasticity. R2 values range from 0 to 1.0, with higher values indicating better skin elasticity. Measurements were collected under standardized conditions at Baseline (Day 0), Week 8, Week 12, and Week 16.
Time Frame: Baseline, Week 8, Week 12, Week 16
Population: 28 participants were assessed at Baseline and Week 8. One participant was lost to follow-up after Week 8, resulting in 27 participants at Weeks 12 and 16. Skin elasticity was measured using the R2 parameter from Cutometer readings at each time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: face
Arm/Group | Epidermal Growth Factor Serum Application
Number analyzed (Participants) | 28
Number analyzed (face) | 28
units on a scale
  Baseline | 0.596 (0.016)
  8 wk | 0.596 (0.013)
  12 wk: number analyzed (Participants) | 27
  12 wk: number analyzed (face) | 27
  12 wk | 0.584 (0.012)
  16 wk: number analyzed (Participants) | 27
  16 wk: number analyzed (face) | 27
  16 wk | 0.553 (0.014)
Statistical Analysis 1: Comparison: Epidermal Growth Factor Serum Application; The statistical analysis utilized repeated measures ANOVA to evaluate changes in facial skin elasticity (R2 parameter) across multiple time points (Baseline, Week 8, Week 12, and Week 16) within the same participants. This approach accounts for the correlation of repeated measures over time; Test type: Superiority — The chosen test was designed to assess whether application of the intervention resulted in any statistically significant differences over time in the primary outcome measure, assuming superiority; p = 0.169, ANOVA — The pre-specified significance threshold was set at p < 0.05. No adjustments for multiple comparisons were applied; Sphericity tested; Greenhouse-Geisser applied if needed. Repeated measures ANOVA accounted for within-subject correlations; Mean Difference (Final Values) = -0.043 — The estimation parameter reflects the change in the R2 elasticity measure from baseline to 16 weeks. The direction of change is based on the final minus baseline value, with baseline serving as the reference point

4. Primary Outcome: Facial Skin Wrinkles
Description: Visioscan measurements were taken at baseline, then at 8, 12, and 16 weeks by using a 4-grade percentage wrinkle improvement scale.
Time Frame: 4 months
Population: The analysis population for this study on facial skin wrinkles using Visioscan included 28 subjects, assessed at Day 0 (baseline), Week 8, Week 12, and Week 16. One subject dropped out at Week 12 and another at Week 16, leaving data from 27 participants for Weeks 12 and 16. Wrinkle improvement was assessed on a 4-grade scale: Grade 1 (0-25%) = slight, Grade 2 (25-50%) = moderate, Grade 3 (50-75%) = marked, Grade 4 (>75%) = significant. Data are presented as mean grades with standard deviation.
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: face
Arm/Group | Epidermal Growth Factor Serum Application
Number analyzed (Participants) | 28
Number analyzed (face) | 28
units on a scale
  baseline | 1 (0)
  8 wk | 1 (0)
  12 wk: number analyzed (face) | 27
  12 wk | 1 (0)
  16 wk: number analyzed (face) | 27
  16 wk | 1 (0)
Statistical Analysis 1: Comparison: Epidermal Growth Factor Serum Application; Test type: Superiority — This study aimed to evaluate changes in wrinkle scores using a 4-grade percentage wrinkle improvement scale across different time points, including baseline, 8 weeks, 12 weeks, and 16 weeks; p = 1.000, ANOVA; Mean Difference (Final Values) = 1 — The Mean Difference represents the change in wrinkle scores from baseline (Day 0) to follow-up at Week 8, Week 12, or Week 16. For example, a Mean Difference of 1.0 indicates a 1-point improvement from baseline to Week 16 (Week 16 - baseline score)

5. Primary Outcome: Facial Melanin Index
Description: Facial pigmentation was assessed using the Mexameter, which measures melanin content via light absorption and reflection. The device reports values on a scale from 0 to 999, where higher values represent greater melanin concentration. Measurements were collected at standardized facial sites at Baseline, Week 8, Week 12, and Week 16. Higher scores indicate worse pigmentation.
Time Frame: 4 months
Population: The analysis population for this study on facial skin pigmentation utilizing Mexameter measurements comprised a total of 28 initially recruited subjects. These participants were assessed at four distinct time points: day 0 (baseline), 8 weeks, 12 weeks, and 16 weeks. One subject loss follow-up at week 12 and week 16.
Measure: Mean (Standard Deviation); unit: unitless index
Units Other Than Participants: face
Arm/Group | Epidermal Growth Factor Serum Application
Number analyzed (Participants) | 28
Number analyzed (face) | 28
unitless index
  Baseline | 244.118 (10.186)
  8 weeks | 246.296 (8.955)
  12 weeks: number analyzed (face) | 27
  12 weeks | 243.605 (10.074)
  16 weeks: number analyzed (face) | 27
  16 weeks | 240.660 (9.838)
Statistical Analysis 1: Comparison: Epidermal Growth Factor Serum Application; The statistical analysis assessed changes in facial melanin index after serum application using repeated measures ANOVA. This method evaluated differences across multiple time points (Baseline, Week 8, Week 12, and Week 16) within the same participants, accounting for the correlated nature of repeated measures; Test type: Superiority — Repeated measures ANOVA was used to detect any change in facial melanin levels due to the intervention; p = 1.000, ANOVA — The p-value indicates no statistically significant change in facial melanin index over time. The p-value was not adjusted for multiple comparisons. Statistical significance was pre-specified at p < 0.05; Sphericity assumptions were checked and addressed as needed (e.g., Greenhouse-Geisser correction); Mean Difference (Final Values) = -3.458 — The estimation parameter reflects the mean change in melanin index from baseline to week 16. Baseline was used as the reference point in the analysis

6. Primary Outcome: Overall Facial Skin Appearance (Photo Evaluation Using SGAIS)
Description: Facial skin appearance was evaluated using the Subject Global Aesthetic Improvement Scale (SGAIS), a 5-point scale where higher scores indicate greater improvement. Scores were assigned by two board-certified dermatologists who assessed photographs taken by the Visia-CR imaging system at Baseline, Week 8, Week 12, and Week 16.
  SGAIS scoring definition:
  1 = Worse, 2 = Mild improvement (<25%), 3 = Moderate (25-49%), 4 = Much improved (50-74%), 5 = Very much improved (≥75%).
Time Frame: 4 months
Population: The analysis population included 28 subjects assessed at baseline, 8, 12, and 16 weeks. One participant was lost to follow-up after week 12.
Measure: Count of Participants; unit: Participants
Arm/Group | Epidermal Growth Factor Serum Application
Number analyzed (Participants) | 28
Participants
  8 weeks Doctor 1 : score 1 | 10
  8 weeks Doctor 1 : score 2 | 18
  8 weeks Doctor 1 : score 3 | 0
  8 weeks Doctor 1 : score 4 | 0
  8 weeks Doctor 2 : score 1 | 12
  8 weeks Doctor 2 : score 2 | 16
  8 weeks Doctor 2 : score 3 | 0
  8 weeks Doctor 2 : score 4 | 0
  12 weeks Doctor 1 : score 1: number analyzed (Participants) | 27
  12 weeks Doctor 1 : score 1 | 5
  12 weeks Doctor 1 : score 2: number analyzed (Participants) | 27
  12 weeks Doctor 1 : score 2 | 20
  12 weeks Doctor 1 : score 3: number analyzed (Participants) | 27
  12 weeks Doctor 1 : score 3 | 2
  12 weeks Doctor 1 : score 4: number analyzed (Participants) | 27
  12 weeks Doctor 1 : score 4 | 0
  12 weeks Doctor 2 : score 1: number analyzed (Participants) | 27
  12 weeks Doctor 2 : score 1 | 11
  12 weeks Doctor 2 : score 2: number analyzed (Participants) | 27
  12 weeks Doctor 2 : score 2 | 14
  12 weeks Doctor 2 : score 3: number analyzed (Participants) | 27
  12 weeks Doctor 2 : score 3 | 2
  12 weeks Doctor 2 : score 4: number analyzed (Participants) | 27
  12 weeks Doctor 2 : score 4 | 0
  16 weeks Doctor 1 : score 1: number analyzed (Participants) | 27
  16 weeks Doctor 1 : score 1 | 5
  16 weeks Doctor 1 : score 2: number analyzed (Participants) | 27
  16 weeks Doctor 1 : score 2 | 12
  16 weeks Doctor 1 : score 3: number analyzed (Participants) | 27
  16 weeks Doctor 1 : score 3 | 9
  16 weeks Doctor 1 : score 4: number analyzed (Participants) | 27
  16 weeks Doctor 1 : score 4 | 1
  16 weeks Doctor 2 : score 1: number analyzed (Participants) | 27
  16 weeks Doctor 2 : score 1 | 10
  16 weeks Doctor 2 : score 2: number analyzed (Participants) | 27
  16 weeks Doctor 2 : score 2 | 12
  16 weeks Doctor 2 : score 3: number analyzed (Participants) | 27
  16 weeks Doctor 2 : score 3 | 5
  16 weeks Doctor 2 : score 4: number analyzed (Participants) | 27
  16 weeks Doctor 2 : score 4 | 0
Statistical Analysis 1: Comparison: Epidermal Growth Factor Serum Application; Improvement in facial appearance was assessed using the Subject Global Aesthetic Improvement Scale (SGAIS), rated independently by two board-certified dermatologists at multiple time points (8, 12, and 16 weeks); Test type: Superiority — A descriptive analysis was performed. No hypothesis testing or power calculation was conducted for this outcome; p = 1.000, Descriptive — The p-value reflects descriptive analysis of SGAIS improvement scores; no statistical testing for significance was conducted; The evaluation involved categorical SGAIS ratings assigned by two independent dermatologists; percentage of participants at week 16 = 44 — This estimate reflects the proportion of participants rated as showing mild improvement on the SGAIS at Week 16, as detailed in the tabular data

7. Secondary Outcome: Subject Satisfaction in Improving Skin Hydration, Elasticity, Wrinkles, and Pigmentation
Description: Using a quartile grading system, (0 = unsatisfied), (1 = slightly satisfied), (2 = satisfied), and (3 = very satisfied)
Time Frame: 4 months
Population: The assessment of participant satisfaction post-treatment involves all twenty-eight participants, with evaluations at 2, 3, and 4 months using a quartile grading system (0 = unsatisfied, 1 = slightly satisfied, 2 = satisfied, 3 = very satisfied). It is important to note that one subject was lost to follow-up since the 12-week mark.
Measure: Count of Participants; unit: Participants
Arm/Group | Epidermal Growth Factor Serum Application
Number analyzed (Participants) | 28
Participants
  8 weeks : very satisfied | 10
  8 weeks : satisfied | 18
  8 weeks : slightly satisfied | 0
  8 weeks : unsatisfied | 0
  8 weeks : NA (loss follow up) | 0
  12 weeks : very satisfied | 5
  12 weeks : satisfied | 21
  12 weeks : slightly satisfied | 1
  12 weeks : unsatisfied | 0
  12 weeks : NA (loss follow up) | 1
  16 weeks : very satisfied | 6
  16 weeks : satisfied | 21
  16 weeks : slightly satisfied | 0
  16 weeks : unsatisfied | 0
  16 weeks : NA (loss follow up) | 1
Statistical Analysis 1: Comparison: Epidermal Growth Factor Serum Application; Satisfaction was assessed at weeks 8, 12, and 16 using a quartile scale: 0 = Unsatisfied, 1 = Slightly satisfied, 2 = Satisfied, 3 = Very satisfied. One participant was lost to follow-up after week 12; Test type: Superiority — Descriptive summary statistics were used to report satisfaction at multiple time points. No inferential testing was performed; Descriptive; No formal statistical hypothesis testing was performed; percentage of participants at week 16 = 75 — The estimated percentage reflects participants who reported a satisfaction score of 2 or 3 at week 16

8. Secondary Outcome: Adverse Events
Description: Adverse events were systematically monitored at 2, 4, 8, 12, and 16 weeks post-treatment initiation.
Time Frame: 4 months
Population: The comprehensive evaluation encompassed a total of 28 subjects. One participant was lost to follow-up at the 12-week mark. Adverse events were systematically monitored through video calls at 2 and 4 weeks post-treatment initiation. On-site evaluations were conducted at 8, 12, and 16 weeks. At each time point, the number of participants analyzed was 28, with one participant lost to follow-up at the 12-week and 16-week evaluations.
Measure: Count of Participants; unit: Participants
Arm/Group | Epidermal Growth Factor Serum Application
Number analyzed (Participants) | 28
Participants
  2 weeks : No adverse event | 28
  2 weeks : Yes adverse event | 0
  2 weeks : Data missing | 0
  4 weeks : No adverse event | 28
  4 weeks : Yes adverse event | 0
  4 weeks :Data missing | 0
  8 weeks : No adverse event | 28
  8 weeks : Yes adverse event | 0
  8 weeks : Data missing | 0
  12 weeks : No adverse event | 27
  12 weeks : Yes adverse event | 0
  12 weeks : Data missing | 1
  16 weeks : No adverse event | 27
  16 weeks : Yes adverse event | 0
  16 weeks : Data missing | 1
Statistical Analysis 1: Comparison: Epidermal Growth Factor Serum Application; The analysis population includes 28 participants. One subject was lost to follow-up at week 12. Adverse events were assessed through video calls at weeks 2 and 4, and in-person visits at 2, 3, and 4 months; Test type: Superiority — This was a descriptive safety analysis. No inferential hypothesis testing was conducted; Descriptive; No formal statistical test was conducted; Percentage adverse events by week 16 = 0 — Descriptive summaries of adverse event incidence are reported in the results tables

ADVERSE EVENTS:
Time Frame: Baseline, Week 8, Week 12, Week 16
Description: Adverse events, including erythema, edema, hyperpigmentation, skin infection, itching, irritation, burning sensation, papules, and acne, were monitored at multiple time points. No adverse events were reported. All 28 enrolled participants were monitored for adverse events, and therefore the Total Number of Participants at Risk is 28 across all adverse event tables.
Arm/Group | Epidermal Growth Factor Serum Application
All-Cause Mortality (participants affected / at risk) | 0/28
Serious Adverse Events (participants affected / at risk) | 0/28
Other Adverse Events (participants affected / at risk) | 0/28

LIMITATIONS AND CAVEATS:
The small sample size should be considered. Further research involving a larger population or control group is recommended for conclusive insights into the efficacy of EGF serum.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-04-10): https://cdn.clinicaltrials.gov/large-docs/89/NCT05724589/Prot_SAP_001.pdf